CLINICAL TRIAL: NCT06498726
Title: Role of Transcranial Doppler and Magnetic Resonance Angiography for Future Management of Sickle Cell Anemia CNS.
Status: Not yet recruiting | Type: Observational
Sponsor: Eman Abdul-Hai (Other)
Responsible Party: Sponsor-Investigator, Eman Abdul-Hai, Assiut, Assiut University
Organization: Assiut University (Other)
Other Study IDs: sickle cell anemia
Record Dates: First submitted 2024-07-07; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Blood Disease; Brain Injuries
MeSH Terms: conditions — Hematologic Diseases; Brain Injuries | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This prospective cross-sectional will include 18 patients who are diagnosed with sickle cell anemia of either sex aged 1 to 18 years old; free from neurological disorders.
  Interventions: Device: transcranial doppler

INTERVENTIONS:
Device: transcranial doppler — Demographic and procedural variables will be extracted from medical record assistants , and analysis of recorded images TCD, MRA ,interpretation reports will be assessed , Completeness of protocol components will be assessed Data accuracy and protocol fidelity will be ensured through site monitoring
  Other Names: MRA

SUMMARY:
This study aimed to determine the Predictive Value of Transcranial Doppler and Magnetic Resonance Angiography for Future Management of Sickle Cell Anemia.

Specific aims are:

Demonstrate silent parenchymal and vascular brain changes that are incidentally observed in neurologically free SCD children using screening TCD and MRA in Pediatric Hematology unit at Assiut University Hospital

Detect any abnormality with vasculopathy, arterial occlusion and old SCI. Strokes in children with SCD can be prevented by checking a transcranial Doppler (TCD) ultrasound,MRA and providing blood transfusions to children with abnormal blood flow on the TCD and detect Silent cerebral and cerebrovascular changes in SCD.

DETAILED DESCRIPTION:
Cerebro-vascular accident is a destructive complication of sickle cell disease, CVA is a important cause of morbidity and mortality individuals with SCD, which cause motor and neurocognitive complications. The CVA pathophysiology can be described by vasculopathy and obstruction caused by the sickle erythrocytes with narrowing of cerebral vessels of the circle of Willis (middle cerebral artery, anterior cerebral artery, anterior communicating artery, internal carotid artery, posterior cerebral artery, and posterior communicating artery).

Patients with sickle cell disease develop vasculopathy and obstruction at specific sites as distal internal carotid artery (ICA) and the proximal segments of the middle cerebral artery (MCA) and anterior cerebral artery (ACA). This Study have been concerned to identify synchronous risk factors for Cerebro-vascular accident and the presence of increase in cerebral blood flow velocity (CBFV) in arterial parts of the polygon of Willis by transcranial doppler (TCD) has been confirmed as the important risk factor for the development of ischemic Cerebrovascular accidents in children and adolescents with SCA. TCD can detect intracranial arterial narrowing caused by arterial vasculopathy associated with SCA. TCD is a non-invasive, portable, and relatively inexpensive method that uses specific areas of the skull to access the intracranial arterial circulation and to measure CBFV in the polygon of Willis arteries, magnetic resonance Angiography (MRA), and cerebral angiography are available for cerebrovascular disease diagnosis.(5-8) However, TCD is due to its operator dependent, it has a narrow application area. Cerebrovascular disease indicates a group of disorders that alter the flow of blood in the brain. The brain's functions can be temporarily or permanently impaired as a result of this change in blood flow. Timely diagnosis and treatment can restore the brain-impaired functions, resulting in a much-improved prognosis for the patients. This review summarizes the basic principles underlying the TCD imaging technique and its utility as a diagnostic tool for cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* (1) age, from 24 months to 18 years; (2) hemoglobinopathy diagnosis of Hb SS; (3) the desire and ability to be screened as evidenced by signed parental informed consent and child's assent; (4) the availability for follow-up for at least 2 years.

Exclusion Criteria:

- 1.Other sickle cell syndromes were excluded because they had a lower or uncertain risk of stroke.

2.A child was excluded from TCD screening for any of the following: an indication for chronic blood transfusion or a contraindication to chronic transfusion, participation in any study involving treatments which might confound the interpretation of the results of the proposed work

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This prospective cross-sectional will include 18 patients who are diagnosed with sickle cell anemia of either sex aged 1 to 18 years old; free from neurological disorders ,at Assiut University pediatric Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
silent parenchymal and vascular brain changes in Sickle cell disease. | TWO YEARS
  the main outcome variable which is to demonstrate silent parenchymal and vascular brain changes that are incidentally observed in neurologically free SCD children using screening TCD and MRA

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deus-Silva L, Bonilha L, Damasceno BP, Costa AL, Yasuda CL, Costa FF, Santos AO, Etchebehere EC, Oquendo-Nogueira R, Fockink R, de Freitas CF, Camargo EE, Li LM, Cendes F, Saad ST. Brain Perfusion Impairment in Neurologically Asymptomatic Adult Patients with Sickle-Cell Disease Shown by Voxel-Based Analysis of SPECT Images. Front Neurol. 2013 Dec 20;4:207. doi: 10.3389/fneur.2013.00207. eCollection 2013. PMID 24391625
- [Background] Helton KJ, Adams RJ, Kesler KL, Lockhart A, Aygun B, Driscoll C, Heeney MM, Jackson SM, Krishnamurti L, Miller ST, Sarnaik SA, Schultz WH, Ware RE; SWiTCH Investigators. Magnetic resonance imaging/angiography and transcranial Doppler velocities in sickle cell anemia: results from the SWiTCH trial. Blood. 2014 Aug 7;124(6):891-8. doi: 10.1182/blood-2013-12-545186. Epub 2014 Jun 9. PMID 24914136